CLINICAL TRIAL: NCT01000402
Title: Assessment and Follow Up Study of Children and Adolescent With Bipolar Disorder
Brief Title: Juvenile Bipolar Disorder Outpatient Program
Acronym: ProCAB
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Luis Augusto Paim Rohde, Federal University of Rio Grande do Sul
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 07-641
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2009-10-23 (Estimated); Status verified 2009-10

CONDITIONS: Bipolar Disorder; Attention Deficit Disorder With Hyperactivity
Keywords: Bipolar Disorder; Attention-Deficit/Hyperactivity Disorder; Genetics; Environmental Factors; Family Factors
MeSH Terms: conditions — Bipolar Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Psychopharmacotherapy (Other): No specific arms; Treatment decision based on available guidelines
  Interventions: Drug: Psychopharmacotherapy

INTERVENTIONS:
Drug: Psychopharmacotherapy — Lithium (according to response, serum levels, and tolerance) 150-1500mg Valproate (according to response, serum levels, and tolerance) 125-2000mg Risperidone (according to response, and tolerance)0.5-6mg Olanzapine(according to response, and tolerance)2.5-20mg Ziprasidone(according to response, and tolerance)40-160mg Topiramate (according to response, and tolerance)25-300mg Quetiapine (according to response, and tolerance)25-500mg Aripiprazole (according to response, and tolerance)5-20mg Lamotrigine (according to response, and tolerance)25-200mg Fluoxetine (according to response, and tolerance) 1-40mg Sertraline (according to response, and tolerance)25-200mg Methylphenidate (according to weight, response, and tolerance)0.3 -0.7mg/kg/day

SUMMARY:
This is an outpatient program for children and adolescents with bipolar disorders. The naturalistic approach of the program will allow a proper investigation of the disorder, assessment of environmental and biological factors, the conduction of treatment studies, and follow-up of the subjects.

DETAILED DESCRIPTION:
Inclusion criteria:

Age 6-17 years old, male and female. Bipolar Disorder I, II, and NOS (subjects presenting episodes of distinct abnormally and persistently elevated, expansive, or irritable mood, accompanied by at least three -or four if the mood is only irritable - Criteria B symptoms and present to a significant degree for at least 24 hours.

Severe Mood Dysregulation (SMD), as defined by Brotman et al. (American Journal of Psychiatry, 2007)

Exclusion criteria:

Presence of a diagnosis of Pervasive Developmental Disorder, Schizophrenia, Drug Use Disorder, and any other counter indications to outpatient treatment (significant suicide or homicide risk)

Diagnosis:

K-SADS-PL-W WASI Clinical Interview

Outcome Measures:

CBCL for general psychopathology YMRS, CMRS-P, CMRS-T for manic symptoms CDRS and CDI for depressive symptoms SNAP-IV for ADHD symptoms Scared-C and Scared-P for anxiety symptoms CGI for clinical impression, CGAS for global functioning Petersen Pubertal Scale Mood Symptom Questionnaire for SMD Screening tests for leaning disorders Family Environmental Scale, Life Events Scale, Expressed Emotion Adjective Checklist, Resilience Scale, Quality of Life for environmental and psychological factors Medication Adverse Events Checklist

ELIGIBILITY:
Inclusion Criteria:

* 6-18 years-old;
* Bipolar Disorder I, II or NOS
* Severe Mood Dysregulation

Exclusion Criteria:

* Schizophrenia
* Pervasive Developmental Disorder
* Drug use disorder
* Severe suicidal or homicidal risk, counterindicating outpatient treatment

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-02; Primary Completion 2012-10 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Changes in manic and depressive symptoms over time using YMRS, CMRS-P, CDRS, and CDI | Naturalistic Study - 2-year follow-up
Polymorphisms at candidate genes for Bipolar Disorder and Attention-Deficit/Hyperactivity Disorder | Naturalistic 2-year follow-up

SECONDARY OUTCOMES:
Changes in ADHD symptoms according to SNAP-IV | Naturalistic 2-year follow-up
Changes in Anxiety symptoms according to the SCARED-C and SCARED-P | Naturalistic 2-year follow-up
Changes in family functioning according to the FES-R, individual functioning according to the EEAC and Resilience Scale, environmental factors according to the Stressful Life Events Scale | Naturalistic 2-year follow-up
Presence and onset of adverse events secondary to treatment | Naturalistic 2-year follow-up
Changes in SMD symptoms according to the Mood Symptom Questionnaire | Naturalistic 2-year follow-up
Changes in general functioning according to the CGI and the CGAS | Naturalistic 2-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Rohde, D.Sc., Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- See also: Official Website of the ProCAB Outpatient Program — http://www.ufrgs.br/procab